CLINICAL TRIAL: NCT06156631
Title: An Evaluation of Newly Developed Multimodal Health Intervention Among Uncontrolled Hypertensive Jordanian Adults in Primary Health Care Setting
Brief Title: Uncontrolled Hypertension Management Among Jordanian Adults
Acronym: DASH-ExMAMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, NASIR AS'AD IBRAHIM MATANI, PhD student, Universiti Sains Malaysia
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NM2991969
Record Dates: First submitted 2023-11-19; First posted 2023-12-05 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Hypertension; Physical Activity; Dietary Habits; Medication Adherence; Motivational Interviewing
MeSH Terms: conditions — Hypertension; Motor Activity; Feeding Behavior; Medication Adherence | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: A Quasi-experimental design will be used to test the efficacy of the intervention (DASH-ExMAMI) on participants. The participants will be allocated into experimental and control groups. The experimental group will complete dietary, physical activity, medication adherence, and anthropometric assessments before and after the intended intervention. Similarly, the control group will be subjected to dietary, physical activity, medication adherence, and anthropometric assessments before and after the intervention, as in the experimental group but receiving only a usual care (UC) as provided by the PHC. The intervention (DASH-ExMAMI) will last ten weeks (ten sessions) and will include DASH dietary instruction and meal planning, self-monitored brisk walking exercise, and a medication adherence intervention based on an individual MI counselling approach.
Who Masked: Outcomes Assessor
Masking Description: A single-blind method will be used for the main outcome measure (BP) in this study. Blood pressure and the anthropometric measurements (height, weight, and waist circumference) will be assessed by a research assistant who doesn't know which group a participant belongs to. However, an open-label method will be applied for the other outcome measures: dietary habits, physical activity, and medication adherence.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants receive DASH-ExMAMI intervention. (Experimental): Jordanian participants who are adults (age between ≥ 18 and 65 years), have had diagnosed with hypertension and has started his or her treatment plan, and have uncontrolled hypertension (The average systolic blood pressure reading that is equal to or higher than 130 mmHg and/or diastolic blood pressure that is equal to or higher than 90 mmHg for the last two patients' records available at the health centre.
  Interventions: Behavioral: DASH-ExMAMI
- Participants who do not receive DASH-Ex MAMI (No Intervention): Jordanian participants who are adults (age between ≥ 18 and 65 years), have had diagnosed with hypertension and has started his or her treatment plan, and have uncontrolled hypertension (The average systolic blood pressure reading that is equal to or higher than 130 mmHg and/or diastolic blood pressure that is equal to or higher than 90 mmHg for the last two patients' records available at the health centre.

INTERVENTIONS:
Behavioral: DASH-ExMAMI — The DASH-ExMAMI consists of ten counseling and health education sessions that each last from 20 to 60 minutes over 10 weeks. The DASH domain will address the following subjects: getting started on DASH, making the move to DASH, tips to reduce salt and sodium, and a week with the DASH eating plan. The Exercise component consists of brisk walking for 30 minutes every day, five days a week. The medication adherence domain is based on the participant's Hill-Bone Compliance to High Blood Pressure Therapy Scale items and their scores. All domains of the intervention are stages and processes of change-matched ones and are provided through 10 motivational interviewing and counseling sessions.
  Other Names: Dietary approach to stop hypertension, exercise and medication adherence behavioral change
  Arms: Participants receive DASH-ExMAMI intervention.

SUMMARY:
This study will evaluate a newly developed multimodal health intervention including dietary approach to stop hypertension (DASH) diet, exercise (Ex), and medication adherence (MA) using motivational interviewing (MI) counselling (DASH-Ex MAMI) for hypertensive Jordanian adults in primary care settings.

DETAILED DESCRIPTION:
This interventional study specifically aims to:

1. Develop a valid multimodal health intervention that includes DASH, exercise, and medication adherence using MI counselling (DASH-ExMAMI) for hypertensive Jordanian adults in primary care settings.
2. Evaluate the effectiveness of the DASH-ExMAMI intervention on systolic and diastolic blood pressure in adults with uncontrolled hypertension in Jordan.
3. Evaluate the effectiveness of the DASH-ExMAMI intervention on the dietary habits scores in adults with uncontrolled hypertension in Jordan.
4. Evaluate the effectiveness of the DASH-ExMAMI intervention on the physical activity scores in adults with uncontrolled hypertension in Jordan.
5. Evaluate the effectiveness of the DASH-ExMAMI intervention on medication adherence scores in adults with uncontrolled hypertension in Jordan.
6. Evaluate the impact of the DASH-ExMAMI intervention on body mass indices (BMI) and waist circumferences (WC) in adults with uncontrolled hypertension in Jordan

ELIGIBILITY:
Inclusion Criteria:

1. Patient's age between ≥ 18 and 65 years old.
2. Has had diagnosed with hypertension and has started his or her treatment plan.
3. Has uncontrolled hypertension: The average systolic blood pressure reading that is equal to or higher than 130 mmHg and/or diastolic blood pressure that is equal to or higher than 90 mmHg for the last two patients' records available at the health center.
4. Has no other comorbidities that contraindicate exercise or restrict DASH diet.
5. Written medical authorization (documented in patient's medical record) by the attending primary healthcare physician approving the patient's participation.

Exclusion Criteria:

1. Pregnant and postpartum women
2. Has severe hypertension (SBP≥ 200 or DBP ≥110). Resting SBP greater than 200mm Hg or DBP greater than 110mm Hg is a relative contraindication to exercise stress testing.
3. Has history of cardio-pulmonary, renal, or musculoskeletal comorbidities that contraindicate exercise or DASH diet.
4. This research will exclude all clients who are contraindicated to undergo treadmill tests with extra precautions: history of myocardial infarction within six months, angina, cardiac dysrhythmias, symptomatic aortic stenosis, and heart failure, pulmonary embolus, infarction or hypertension, myocarditis or pericarditis, or endocarditis, aortic dissection, history of renal impairment, brittle diabetes mellitus, bronchial asthma, musculoskeletal problems that might worsen by exercise, and mental health problems that interfere with the comprehension of the intervention and its related safety measures. Clients with a history of metabolic disorders and who follow a specific diet restriction will also be excluded such as celiac disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2024-06-07 (Actual); Primary Completion 2024-09-05 (Actual); Study Completion 2024-10-07 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure (SBP) | At two points: pre-intervention (baseline) and post-intervention (after 10 weeks)
  the average measurement of systolic blood pressure in mmHg using valid automated blood pressure apparatus.
Diastolic blood pressure (DBP) | At two points: pre-intervention (baseline) and post-intervention (after 10 weeks)
  the average measurement of diastolic blood pressure in mmHg using valid automated blood pressure apparatus.

SECONDARY OUTCOMES:
Dietary habits | At two points: pre-intervention (baseline) and post-intervention (after 10 weeks)
  The scores obtained by the 'start the conversation- food frequency questionnaire ' STC-FFQ' which quantifies healthy and unhealthy food components consumed by the clients for the last week over a few months and gives a specific score for each component, with the summary score ranging from 0 to 16-the lowest score indicating the healthiest eating pattern.
Physical activity | At two points: pre-intervention (baseline) and post-intervention (after 10 weeks)
  The scores obtained by the international physical activity questionnaire -short form IPAQ-SF which inquiries about three distinct types of activity in three domains (leisure time, domestic/gardening, and work and transport-related activity, as well as sitting). Walking, moderate-intensity activities, and vigorous-intensity activities are the specific types of activity that are assessed; frequency (measured in days per week) and duration (minutes per day) are gathered individually for each specific type of activity. The higher the score- expressed in Metabolic Equivalent of Task (MET)-min per week, the more intense the physical activity
Medication adherence | At two points: pre-intervention (baseline) and post-intervention (after 10 weeks)
  The scores obtained by the Hill-Bone Compliance to High Blood Pressure Therapy Scale (HB-HBP) which evaluates patient behaviors in three key areas of high blood pressure treatment: 1) reduced sodium intake, 2) appointment keeping, and 3) medication taking.
Body mass index (BMI) | At two points: pre-intervention (baseline) and post-intervention (after 10 weeks)
  the output measure of dividing participant's weight in kilograms by their height in meters squared, or BMI = weight (in kg)/height2 (in m2).
Waist circumference (WC) | At two points: pre-intervention (baseline) and post-intervention (after 10 weeks)
  The value of WC measurement for a participant at the end of normal breaths, horizontally to the floor level, and at the midpoint between the upper of the iliac crest and the lowest palpable rib in the mid axillary line.

CONTACTS AND LOCATIONS:
Locations (4):
- Jordan (4):
  - Al Barha Health Center, Irbid
  - Al Tattweer Al Hadhary Health Center, Irbid
  - Al Zahrawi Health Center, Irbid
  - Maruw Health Center, Irbid